CLINICAL TRIAL: NCT00595725
Title: Intra-Operative Lymphatic Mapping in Patients With Invasive Carcinoma of the Cervix or Endometrial Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 02-127
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Cervical Cancer; Endometrial Cancer; Cervical Carcinoma
Keywords: Cervix; Endometrium; Cervical Carcinoma; Lymphatic Mapping
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Lymphatic Mapping

INTERVENTIONS:
Other: Lymphatic Mapping — Intra-Operative Lymphatic Mapping

SUMMARY:
The purpose of this study is to learn if a surgical technique called intraoperative lymphatic mapping can accurately identify the lymph node that is at greatest risk if endometrial or cervical cancer spreads to the lymph nodes.

Early cervical cancer is usually treated by removing the cervix, tissue around the cervix, and the upper vagina. If needed, the uterus is also removed. The treatment also includes removing lymph nodes from the pelvis. Endometrial cancer is usually treated by removing the cervix, uterus, fallopian tubes and ovaries.

The treatment also includes removing lymph nodes from the pelvis.

DETAILED DESCRIPTION:
Patients with FIGO stage I endometrial cancer or patients with FIGO stage I-IIA invasive cervical cancer and who will be undergoing surgical management to include a lymphadenectomy.

↓ Injection of radioisotope and preoperative lymphoscintigraphy with Tc99m either the day before or on the day of surgery by the Nuclear Medicine Department.

↓ Intraoperative lymphatic mapping with blue dye and gamma probe.

↓ Hysterectomy, Radical hysterectomy and/or radical trachelectomy and pelvic lymphadenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with endometrial cancer diagnosed on endometrial biopsy or dilatation and curettage.
* Patients with invasive cervical cancer diagnosed on cervical biopsy or cone biopsy.
* Patients with a performance status of 0, 1, 2, or 3 by the Gynecologic Oncology Group criteria (Appendix).
* Patients with stage I to ~IIA invasive cervical cancer disease according to the International Federation of Gynecology and Obstetrics (FIGO) clinical staging criteria (Appendix).
* Patients with clinical stage I endometrial cancer
* Patients who will undergo surgery to include a hysterectomy, radical hysterectomy and/or radical trachelectomy and bilateral lymphadenectomy via laparotomy or laparoscopy
* Patients who have signed an approved informed consent.

Exclusion Criteria:

* Patients with history of prior pelvic or para-aortic lymphadenectomy.
* Patients with stage IIB-IV invasive cervical cancer by FIGO criteria.
* Patients with recurrent endometrial or cervical cancer.
* Patients with prior pelvic radiation.
* Any patient with endometrial or cervical cancer treated with neoadjuvant chemotherapy and radiation therapy.
* Patients with a performance score of 4 by the Gynecologic Oncology Group criteria or who are not good surgical candidates (Appendix).
* Patients with grossly infected primary tumors.
* Patients with known allergy to triphenyl-ethane compounds.
* Patients with known deficiency of Glucose-G-Phosphate Dehydrogenase.
* Patients with known Hemolytic Anemia from Pyruvate Kinase and G6PD Deficiencies.
* Severe Renal Disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2003-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of identifying the sentinel lymph node in patients with endometrial and invasive cervical cancer using a combination of radioisotope and blue dye. | 7 years

SECONDARY OUTCOMES:
To determine the feasibility of locating sentinel nodes in the pelvis and/or paraaortic region with preoperative lymphoscintigraphy. | 7 years
To document the location of the sentinel nodes in patients with invasive cervical cancer. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary Gemignani, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org